CLINICAL TRIAL: NCT01358643
Title: Operation Enduring Freedom and Operation Iraqi Freedom (OEF/OIF) Veteran Preferences for and Feasibility of Automated Physical Activity Interventions: A Pilot Study
Brief Title: Operations Enduring Freedom and Iraqi Freedom (OEF/OIF)Veteran Preferences for Automated Physical Activity Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: VA Ann Arbor Healthcare System (U.S. Federal Agency)
Responsible Party: Caroline Richarson, MD, Va Ann Arbor Healthcare System
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: LIP 41-114
Record Dates: First submitted 2011-05-19; First posted 2011-05-24 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-05

CONDITIONS: Physical Activity
Keywords: OEF/OIF; Physical Activity; Preferences
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- P90X + Sparkpeople (Other): For six weeks of the study participants will use the P90X tools and for the other six weeks participants will use Sparkpeople tools.
  Sparkpeople is a web based diet and exercise program in which the participant can track their diet and exercise progress and read and post messages to a large online community of others who are also trying to lose weight.
  P90X is A DVD based home exercise program that guides the participant through a daily exercise routine.
  Interventions: Other: Three home-based diet and exercise programs
- P90X + BodyMedia Fit (Other): For six weeks participants will use the P90X tools and for the other six weeks participants will use the BodyMedia Fit Device.
  P90X is a DVD based home exercise program that guides the participant through a daily exercise routine.
  BodyMedia Fit is a program in which the participants wears a small device on their arm that measures their physical activity and allows you to upload detailed physical activity data to a web site to help them track your progress.
  Interventions: Other: Three home-based diet and exercise programs
- BodyMedia Fit + Sparkpeople (Other): For six weeks participants will use the BodyMedia Fit devise and for the other six weeks participants will use the Sparkpeople program.
  BodyMedia Fit is a program in which the participants wears a small device on their arm that measures their physical activity and allows you to upload detailed physical activity data to a web site to help them track your progress.
  Sparkpeople is A web based diet and exercise program in which the participant can track their diet and exercise progress and read and post messages to a large online community of others who are also trying to lose weight
  Interventions: Other: Three home-based diet and exercise programs

INTERVENTIONS:
Other: Three home-based diet and exercise programs — All research activities are outpatient. This pilot study will be a crossover study of two 6-week programs. The participant will be involved for 15 weeks.
  Thirty OEF/OIF veterans with BMI > 30 will be recruited to test the diet and exercise programs. Each veteran will test only two of the three programs described above. The participants will use the the programs for six weeks then crossover and use a second program.

SUMMARY:
The purpose of this pilot is to assess the feasibility and potential effectiveness of three specific e-health approaches. One approach, SparkPeople.com, involves the use of social media and can be accessed through a free website. This approach has the potential to provide support through an on-line community as well as a number of diet/weight and physical activity related tools. A mobile phone application is also available for those with smart phones. The second approach, BodyMedia, involves the use of an objective monitoring device that tracks all activity. This information can be uploaded to a website to provide ongoing monitoring and feedback about activity and energy expenditure. The third approach, P90X, involves a DVD based resistance focused exercise program. While DVD programs are not necessarily considered e-health, participants will be encouraged to participate in online community forums associated with the program. All participants, regardless of randomization, will be given 4 point of decision prompts that are laminated 8.5x11 posters encouraging healthier behaviors to display in various areas of their home.

The specific aims are:

1. To assess the effect of the intervention on weight, activity levels, depression, and adherence.
2. To determine level of interest, perceptions, feasibility and satisfaction of the proposed interventions (i.e. SparkPeople.com vs. BodyMedia vs. P90X) with particular attention to: 1) social media; 2) food logs; 3) objective monitoring of physical activity; 4) use of point systems

DETAILED DESCRIPTION:
This is a pilot study designed to better understand what elements/strategies help to engage Operations Enduring Freedom and Iraqi Freedom (OEF/OIF) veterans in an e-health program for promoting weight loss and increasing physical activity. These data will be used as pilot information for a larger study to assess the effectiveness of using an e-health approach to promote weight loss and increase physical activity among post-deployment OEF/OIF veterans who are at risk for developing diabetes. Additionally, we seek to recognize any effects of the intervention on other health-related outcomes, such as stress, depression or other mental health measures, chronic pain, sleep, quality of life, satisfaction with care/ Veteran Affairs Health system, employment status, social support/connectedness.

Post-deployment OEF/OIF veterans worry about gaining weight and believe regular physical activity is beneficial, yet many don't exercise due to health problems and/or chronic pain. Healthy eating combined with physical activity are key strategies in maintaining or losing weight and is important in preventing diabetes, cardiovascular disease and other preventable illnesses as well as managing many mental health conditions and reducing chronic pain symptoms. In addition, maintaining or improving physical activity/exercise may be an effective strategy for addressing other post-deployment issues: stress, social issues.

E-health strategies may be an effective and potentially preferred as well as efficient (cost-effective) way to deliver or assist OEF/OIF veterans with health and lifestyle related health behaviors. There is a growing array of e-health tools, technologies and approaches to assist people with diet-related issues (for weight loss or maintaining a healthy weight) and to encourage physical activity. This includes cell phone applications, objective monitoring devices such as pedometers and web-based programs (as well as combination of these different strategies). However, the most effective and efficient way to encourage healthy eating and weight loss/maintenance or promote physical activity remains an open question and which tools and technologies might best engage the OEF/OIF veteran population in addressing these lifestyle issues is yet to be determined.

OEF/OIF Coordinators will include the study recruitment flyer in their initial informational mailing to new OEF/OIF veterans and publish the flyer in their monthly newsletter. The recruitment flyer will encourage interested veterans to contact study staff via a toll free number (where they will leave a message) or email. During one-on-one meetings, Coordinators will identify overweight and obese OEF/OIF veterans who are interested in losing weight with physical activity and with the veterans permission will forward the veterans name and phone number to the research study staff by leaving a voice mail on the study phone line. During these meetings, the OEF/OIF Coordinators will also provide basic information regarding the program and provide the Veteran a recruitment flyer. Recruitment flyers will also be posted at strategic locations around the VA with the approval of Public Affairs. Should study staff fail to meet recruitment goals through the assistance of the OEF/OIF Coordinators and posted flyers, primary care physicians (PCPs) will also be educated on the study and given study recruitment flyers to give to potentially eligible patients. With the permission of the veteran, PCPs will forward the veterans name and phone number to the research study staff by leaving a voicemail on the study phone line.

Potential participants will be contacted by phone to be screened for eligibility. If eligible, participant will be asked to come to the Ann Arbor Veterans Affairs Healthsystem (VA) for a 1 ½ to 2 hour enrollment session. Patients will be consented at the start of this enrollment visit, prior to the commencement of any research activities.

All research activities are outpatient. This pilot study will be a crossover study of two 6-week programs. The participant will be involved for 15 weeks.

The three home base diet and exercise programs we are testing are:

1. A web based diet and exercise program in which you can track your diet and exercise progress and read and post messages to a large online community of others who are also trying to lose weight. (Sparkpeople.com)
2. A program in which you wear a small device on your arm that measures your physical activity and allows you to upload detailed physical activity data to a web site to help you track your progress. (Bodymedia Fit)
3. A DVD based home exercise program that guides you through a daily exercise routine. (P90X)

Thirty OEF/OIF veterans with body mass index (BMI) > 30 will be recruited to test the diet and exercise programs. Each veteran will test only two of the three programs described above.

Participants will be informed about the study by OEF/OIF coordinators, medical providers or by reading posters about the study posted in outpatient areas in the Ann Arbor VA Medical Center. Contact information for veterans who express an interest and give permission will be forwarded to the research staff. Research staff will call the potential participant on the phone, briefly describe the study and then complete a short eligibility screening questionnaire. Eligible and interested participants will schedule an initial in person study visit.

At the initial study visit, participants will

* Complete the informed consent process and sign an informed consent document.
* Receive instructions for completing an online survey to be completed during the visit or at home
* Have height and weight recorded by the research coordinator
* Be randomly assigned to test two of the three diet and exercise programs described above
* Receive instructions and related equipment or materials for the first program to test.
* Schedule a follow up visit to cross over to the second program after 6 weeks.

Participants will then test the diet and exercise program at home for 6 weeks.

. At this second visit, the cross over visit, participants will

* Return the materials from the first program they tested
* Have weight rechecked
* Receive instructions on filling out a second online survey asking about experience with program 1 to be completed during the visit or at home
* Complete a 30 minute interview or schedule a time to complete the interview by phone
* Receive instructions and related equipment or materials for the second program.

Participants will then test the second program at home for 6 weeks.

Participants will then arrange with the study coordinator to return the equipment and materials for the second intervention tested, complete a third online survey and a second interview.

Participants may choose to complete the study without a third VA visit. They would return equipment and materials by mail at the VA's expense, complete the final survey online from home and complete the final interview by phone. Study staff will ask participant for self-reported weight measurement if the final visit is done remotely. For participants who do come to the VA for the final assessment, we will also recheck their weight.

Study staff may contact participants by email or phone to remind participants to complete surveys, upcoming phone interviews, and upcoming research visits. If participant does not complete survey online, study staff will offer to mail the survey for participant to complete at home (including a return envelope), or doing the survey by phone.

If participants test the SparkPeople.com website, they will receive an email from study staff with video clips that describe the website in further detail. The will also receive emails directly from Sparkpeople.com depending on how they set their profile.

If participants test the BodyMedia fit device, BodyMedia will send an email directly to the participant with directions on setting up their account.

All three of the diet and exercise programs we are testing in this study are commercially available home exercise programs and they are not programs developed by or delivered by the VA or VA staff.

Please note: At initial study visit, participant is randomized to 2 of the 3 possible interventions.

* The BodyMedia Fit device has nickel contacts on the device. These contacts will be directly next to skin. If participant has known nickel allergy and randomized to BodyMedia Fit group, they will not participate in Body Media Fit intervention. Participant will be given the intervention they were not selected for and given necessary instructions.
* If participant has an unknown nickel allergy and they have a reaction to the BodyMedia Fit device, study staff will document in file on I: drive and tell the participant to stop wearing the device. The participant will wait until the end of the 6 weeks without an intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Identified as an Operations Enduring Freedom and Iraqi Freedom (OEF/OIF) veteran;
2. BMI of 30 or greater;
3. Able to walk at least one block without stopping;
4. Access to a computer on a daily basis with an available USB (universal serial bus) port with high-speed Internet access;
5. Have a working email address;
6. Have a working DVD player to view standard DVDs;
7. be able to communicate in English.

Exclusion Criteria:

1. Currently pregnant;
2. Cannot walk at least one block;
3. Have been referred to the ASPIRE program or are participating in the ASIPRE program;
4. Have dial-up internet access only;
5. Any medical condition that might make it dangerous or medically inappropriate to engage in a diet and exercise program as deemed by the study physician.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Perceptions of Operations Enduring Freedom and Iraqi Freedom (OEF/OIF) Veterans of Different Physical Activity Interventions: Change from Baseline in perceptions of physical activity at 6 weeks and 12 weeks | 6 weeks, 12 weeks
  Perceptions of OEF/OIF Veterans of different physical activity interventions in an e-health program for promoting weight loss and increasing physical activity are the main outcome. Change from Baseline in perceptions of physical activity at 6 weeks and 12 weeks will be measured. These data will be used as pilot information for a larger study to assess the effectiveness of using an e-health approach to promote weight loss and increase physical activity among post-deployment Operations Enduring Freedom and Iraqi Freedom (OEF/OIF) veterans who are at risk for developing diabetes.

SECONDARY OUTCOMES:
Other health-related outcomes: Change from Baseline in health-related outcomes at 6 weeks and 12 weeks | 6 weeks, 12 weeks
  Additionally, we seek to recognize any effects of the intervention on other health-related outcomes, such as stress, depression or other mental health measures, chronic pain, sleep, quality of life, satisfaction with care/Veteran Affairs Healthsystem, employment status, social support/connectedness. Change from Baseline in health-related outcomes (mentioned above) at 6 weeks and 12 weeks will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Richardson, MD, Principal Investigator — VA Ann Arbor Healthcare System
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, Michigan, United States